CLINICAL TRIAL: NCT04716153
Title: Impact of a Sensory Rehabilitation Program on Olfactory-gustatory Alterations in Patients Treated With Chemotherapy for Haematological Cancer
Acronym: RE-NEZ-SENS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolement difficulties
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL20_0187
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Olfactivo-gustatory Disorder; Lymphoma; Haematological Cancer
Keywords: sensory rehabilitation; autograft autologous stem cell transplantation; multiple myeloma; chemotherapy; taste, smell; quality of life; nutrition; lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Anosmia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Ramdonized, controlled study with 2 parallel arms (interventional and control). Patients in the interventional arm will follow a multi-factor sensory rehabilitation program focused on smell and taste with daily use (3 times a day) of Liposomal sprays (LipoSaliva® : mouth and LipoNasal® : nose) between V0 and V1.
  The control group will only receive the usual care provided for as part of routine care. It consists of a nutritional assessment at home by a dietician, with monitoring of intake and weight, in order to readjust nutritional care.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Patients in the interventional arm will follow a multifactorial sensory rehabilitation program focused on smell and taste that integrates several non-drug interventions, which are part of the current recommendations: program of workshops at the technical center, hydration of the mucous membranes with daily (3 times a day) liposomal sprays (LipoSaliva® and LipoNasal) between V0 and V1, presentation of visual dishes.
  The workshops will take place at the frequency of one session of 2 hours per week and will last for 3 weeks. Each session will accommodate a minimum of 2 participants. The program will include 3 workshops on olfactory rehabilitation and taste rehabilitation.
  Exercises (taking up the themes discussed) will be carried out at home between 2 workshops.
  Interventions: Other: Multifactorial sensory rehabilitation workshops; Other: Tests and Questionnaire
- Control (Other): The control group only receives the usual care provided for as part of routine care. It consists of a nutritional assessment at home by a dietician, with monitoring of intake and weight, in order to readjust nutritional support. A systematic search for oral mycosis is carried out in order to treat.
  The foods that the patient prefers, identified from a list of authorized foods, are preferred or even fortified.
  Patients in the control group will be able to benefit from the rehabilitation workshops if they wish at the end of the study.
  Interventions: Other: Usual care; Other: Tests and Questionnaire

INTERVENTIONS:
Other: Multifactorial sensory rehabilitation workshops — A multifactorial sensory rehabilitation Workshops : a multifactorial program in order to optimize the recovery of flavors, focused on smell and taste which integrates several non-drug interventions, which are part of the current recommendations: hydration of the mucous membranes with daily (3 times a day) liposomal sprays (nose and mouth), presentation of visual dishes.
  Arms: Interventional
Other: Usual care — The control group only receives the usual care provided for as part of routine care. It consists of a nutritional assessment at home by a dietician, with monitoring of intake and weight, in order to readjust nutritional support. A systematic search for oral mycosis is carried out in order to treat.
  The foods that the patient prefers, identified from a list of authorized foods, are preferred or even fortified.
  Arms: Control
Other: Tests and Questionnaire — fulfillment of Taste Strips Test, Sniffin'sticks test and QGO, FACT-G, HADS, l'EVA des ingesta and GPAQ questionnaires to assess the quality of life of patients

SUMMARY:
Proposition of a sensory rehabilitation program that could reduce the olfactory-gustatory alterations in patients who have been treated with chemotherapy for Haematological Cancer, and also improve their life quality, psychological well-being, and nutrition.

DETAILED DESCRIPTION:
Disturbances in taste and smell affect a considerable proportion of patients treated with chemotherapy. In hematology, dysgeusia depends on the type pathology and the treatments themselves. It impacts the quality of life, leads to significant emotional and social consequences, affects the intake, weight and nutritional status of patients.

Olfactory-taste disorders can be assessed using subjective and objective tests. There are no international clinical recommendations for the management of taste and olfactory disturbances associated with chemotherapy in hematological cancers. Also, this study proposes to evaluate a taste and olfaction rehabilitation program based on national standards and recent research. It will help fill gaps in the assessment and management of patients treated for Haematological cancer.

Hypothesis is that this sensory rehabilitation program should make it possible to reduce the olfactory-gustatory changes in patients who have been treated with Chemotherapy for Haematological cancer and significantly improve their quality of life, their psychological well-being and their nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and ≤ 75 years old
* Patient with olfactory or gustatory disorders
* Patient who has completed chemotherapy for haematological cancer

Exclusion Criteria:

* Eating disorder known prior to anti-cancer treatment, bulimic, anorexic or binge eating disorder (DSM-V criteria)
* Refusal to sign the free and informed consent
* Hypersensitivity to one of the components of liposomal sprays (Liposaliva® or liponasal®)
* COVID + patient in the previous 3 months
* Performance status ECOG 3 or 4
* Patient included in another clinical trial modifying taste / olfaction
* Artificial nutrition post-chemotherapy
* Known food allergies
* Having a reading level in French that may interfere with a good understanding of the protocol and the questionnaires
* Presenting visual or hearing deficits uncorrected to normal and which may affect the proper completion of the questionnaires
* Patient under curatorship or tutorship.
* Patient deprived of liberty
* Pregnant or breastfeeding patient
* Not be affiliated with a French social security scheme or beneficiary of such a scheme

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2026-01-14 (Actual); Study Completion 2026-01-14 (Actual)

PRIMARY OUTCOMES:
Assessment of the olfactometry | 3 months
  Evolution of the Score of the "Sniffin'sticks" test from the initial score (V0), which itself includes an olfactory discrimination, olfactory threshold and olfactory identification score (with a cut-off of ≤ 15 for anosmia, ≥ for normonosmia and hypoanosmia for a score between 15 and 30)

SECONDARY OUTCOMES:
Assessment of the gustometry | up to 6 months
  Score in the "Taste Strips" test, Hypoageusia scores being for participants aged 18 to 40, <19 for women and <17 for men; for participants aged 41 to 60, score <15 for women and 9 for men; for participants over 60, score <10.2 for women and <9 for men
Variation of Taste and Smell Survey score | up to 6 months
  Variation of the taste and Smell Survey score
Assessment of the Quality of life | Up to 6 months
  Quality of life scores, obtained on the FACT-G scale. This is a 27-point self-administered questionnaire that measures the quality of life of patients with cancer. The FACT-G measures physical, functional, social / family factors, and emotional well-being as well as physician / patient relationship satisfaction and concerns. All items are rated on a 5-point Likert scale based on the week prior to the assessment.
Assessment of the Psychological distress | u pto 6 months
  The psychological distress score objectified by the Hospital Anxiety Depression Scale (HADS). This self-questionnaire, validated in French, contains 14 items. It is simple, sensitive and specific. It has been validated in cancer patients, that it is rapid (completion time around 5 minutes), and allows the calculation of 2 sub-scores for anxiety and depression in addition to an overall level. Finally, this tool is sensitive to changes both during the course of medical illnesses and in response to psychopharmacological interventions.
Assessment of the physical activity | up to 6 months
  assessed by the score at GPAQ scale (Bull, Maslin, & Armstrong, 2009)
Variation of the patient weight | up to 6 months
  assessed by BMI between the beginning and the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Franciane PAUL, Dr., Study Director — UH of Montpellier
Locations (1):
- Hematology Department, University Hospital Center, Montpellier, France